CLINICAL TRIAL: NCT01099085
Title: Placebo-controlled, Double-blinded Phase III Trial of XP (Capecitabine/CDDP) Simvastatin in Advanced Gastric Cancer Patients
Brief Title: Trial of XP (Capecitabine/CDDP) Simvastatin in Advanced Gastric Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-12-019
Record Dates: First submitted 2010-04-04; First posted 2010-04-06 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Gastric Cancer
Keywords: gastric cancer, unresectable/metastatic
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- XP/simvastatin (Active Comparator): Capecitabine/cisplatin + simvastatin
  Interventions: Drug: Simvastatin
- XP/placebo (Placebo Comparator): Capecitabine/cisplatin + placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — simvastatin 40 mg qd daily
  Arms: XP/simvastatin
Drug: Placebo — Placebo
  Arms: XP/placebo

SUMMARY:
Based on antitumor activity of statin, we designed a phase III study of capecitabine/CDDP chemotherapy plus a low-dose simvastatin that is equivalent to cardiovascular dose in advanced gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically confirmed diagnosis of gastric adenocarcinoma or gastroesophageal junction adenoca (i.e. an adenocarcinoma with > 50% extension in the stomach)
2. patients must present with stage IV disease not amenable to surgery, radiation or combined modality therapy with curative intent. Patients previously undergoing local treatment (surgery and/or radiation) must have subsequently progressed or recurred
3. measurable or evaluable disease according to RECIST
4. age, 18 years or older
5. ECOG performance status 0 - 2
6. adequate organ function as defined by the following criteria absolute neutrophil count (ANC) ≥ 1,500/ul platelets ≥ 100,000/ul AST/ALT ≤ 2.5 x ULN, ≤ 5.0 x ULN if liver involvement Total serum bilirubin ≤ 3.0 mg/dL
7. signed written informed consent

Exclusion Criteria:

1. severe co-morbid illness and/or active infections
2. pregnant or lactating women
3. active CNS metastases not controllable with radiotherapy or corticosteroids
4. active and uncontrollable bleeding from gastrointestinal tract
5. known history of hypersensitivity to study drugs
6. patients who are already on statin treatment for hyperlipidemia control (if ≥ 1 year interval from the last statin dose, the patient is eligible for study entry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival of XP ± simvastatin | 1-year PFS

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Cancer Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim ST, Kang JH, Lee J, Park SH, Park JO, Park YS, Lim HY, Hwang IG, Lee SC, Park KW, Lee HR, Kang WK. Simvastatin plus capecitabine-cisplatin versus placebo plus capecitabine-cisplatin in patients with previously untreated advanced gastric cancer: a double-blind randomised phase 3 study. Eur J Cancer. 2014 Nov;50(16):2822-30. doi: 10.1016/j.ejca.2014.08.005. Epub 2014 Sep 15. PMID 25218337